CLINICAL TRIAL: NCT04986527
Title: Chest Tube Management in Traumatic Pneumothorax: Does Duration of Suction Matter
Brief Title: Duration of Chest Tube Suction in Traumatic Pneumothorax
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study does not have funding
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael J Nabozny, MD, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005364
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24 hours of suction (Active Comparator): Subjects with chest tubes kept to -20 cmH2O suction for 24 hours prior to water seal
  Interventions: Procedure: Chest tube suction
- 48 hours of suction (Experimental): Subjects with chest tubes kept to -20 cmH2O suction for 48 hours prior to water seal
  Interventions: Procedure: Chest tube suction

INTERVENTIONS:
Procedure: Chest tube suction — The chest tubes will be inserted using our institutional standard chest tube insertion tray. The chest tubes used will be our institutional standard and will range from 14 to 32Fr in size. After chest tube placement, an Atrium Oasis Dry Suction Water Seal Chest Drain (Getinge USA Sales, LLC) will be used.

SUMMARY:
The purpose of this pilot study is to determine whether chest tube suction duration, 24 hours vs 48 hours, prior to water seal affects outcome and length of stay after placement for traumatic pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* Trauma service consult/patient
* Traumatic pneumothorax with chest tube placed within 0-24 hours of presentation and confirmation of adequate position
* Age >18
* Blunt or penetrating mechanism
* Chest tubes sizes 14 to 32Fr
* Chest tubes placed by residents on the trauma surgery service supervised by attending trauma surgeons or placed by the attending surgeon themselves
* Presence of single chest tube in one or both pleural cavities (single unilateral or bilateral tubes)
* Subjects with decision making capacity (DMC) who are able to provide written consent. DMC will be determined by the consenting physician through a teach back mechanism. Subjects must demonstrate understanding of the situation, appreciation of the consequences of their decision, reasoning of their thought process, and be able to communicate their wishes.

Exclusion Criteria:

* Age <18
* Pregnant patients
* Prisoners
* Mechanically ventilated in ICU for more than 24 hours while chest tube in place
* Chest tubes placed as part of, or present during, a thoracic operation
* History of surgery involving pleural cavity ipsilateral to chest tube
* Subjects with more than one chest tube on the ipsilateral side at any time prior to study chest tube removal
* Subjects with chylothorax or empyema
* Subjects with chest tubes that are withdrawn or removed unintentionally
* Subjects with known or suspected bronchial injury
* Subjects with bullous emphysema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Chest tube dwell time | up to 1 month
  Total time that chest tube is in place from insertion to removal

SECONDARY OUTCOMES:
Number of participants with reaccumulation of pneumothorax | up to 3 days
  After transition to water seal and stopping suction, incidence of reaccumulation of pneumothorax requiring suction or replacement of chest tube.
Number of participants with at least one pulmonary complications | up to 1 week
  Pulmonary complications are defined as increased oxygen requirements, shortness of breath or unplanned intubations following placement to suction.
Readmission to hospital | 30 days
  Number of participants readmitted to the hospital within 30 days
Transfer to ICU | up to 1 week
  Number of participants with an unplanned transfer to the intensive care unit
Median length of stay | Up to 1 year
  Median length of stay in the hospital after chest tube placement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No